CLINICAL TRIAL: NCT05885958
Title: Timing of Active Void Trials After Urogynecologic Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Simone Fertel, Primary Investigator, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY005629
Record Dates: First submitted 2023-05-22; First posted 2023-06-02 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Postoperative Care; Urinary Catheters; Urogynecology
MeSH Terms: interventions — Time

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate (Experimental): Patients will be given up to 30 minutes to void during the active void trial postoperatively.
  Interventions: Other: Time
- Extended (Experimental): Patients will be given up to 60 minutes to void during the active void trial postoperatively.
  Interventions: Other: Time

INTERVENTIONS:
Other: Time — Patients will be given up to 30 minutes to void.
  Arms: Immediate
Other: Time — Patients will be given up to 60 minutes to void.
  Arms: Extended

SUMMARY:
The goal of this clinical trial is to learn about active void trial pass rates in patients undergoing urogynecologic surgery. The main question it aims to answer is the comparison in pass rate during active void trial between women who are given 30 minutes versus 60 minutes to void following urogynecologic surgery.

Patient will be randomized to two arms prior to scheduled surgery. During the active void trial, women will be allotted up to 30 minutes or up to 60 minutes to void depending on respective randomization.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing a urogynecologic surgery at Tampa General Hospital and who are seen preoperatively at the University of South Florid Urogynecology clinic
* Women undergoing a urogynecologic surgery where a postoperative active void trial is indicated
* Planned for same day surgery
* Women able to consent for themselves
* Speak English and/or Spanish as preferred language

Exclusion Criteria:

* Imprisoned patients
* Females under the age of 18 years old
* Women who are unable or unwilling to consent to participation
* Women who are planning to stay inpatient overnight
* Women with history of urinary retention or neurogenic bladder
* Women undergoing procedure that is not standard of care to perform a void trial (includes sacral neuromodulation, botox to the pelvic floor, cystoscopy with hydrodistension, urethral bulking, etc)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 231 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Pass Rate | 60 minutes
  to compare the active void trial pass rate between arms

SECONDARY OUTCOMES:
Time in PACU | 6 hours
  to compare overall time spent in the PACU between arms
Pass Rate After Failing | 60 minutes
  to assess the overall pass rate of active void trial after failed first attempt
UTI | 2 weeks
  to assess rate of urinary tract infection after surgery
Surgical Procedures Performed Prior to Active Void Trial | 2 years
  to compare types of surgery women are having with the rate of void trial passing

CONTACTS AND LOCATIONS:
Locations (1):
- USF Urogynecology Clinic, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barber MD, Walters MD, Karram MM, et al. Walters & Karram Urogynecology and Reconstructive Pelvic Surgery - E-Book: Elsevier Health Sciences; 2021
- [Background] Lo TS, Shailaja N, Hsieh WC, Uy-Patrimonio MC, Yusoff FM, Ibrahim R. Predictors of voiding dysfunction following extensive vaginal pelvic reconstructive surgery. Int Urogynecol J. 2017 Apr;28(4):575-582. doi: 10.1007/s00192-016-3144-z. Epub 2016 Sep 19. PMID 27647467
- [Background] Kim JW, Moon du G, Shin JH, Bae JH, Lee JG, Oh MM. Predictors of Voiding Dysfunction after Mid-urethral Sling Surgery for Stress Urinary Incontinence. Int Neurourol J. 2012 Mar;16(1):30-6. doi: 10.5213/inj.2012.16.1.30. Epub 2012 Mar 31. PMID 22500251
- [Background] Mills JT, Rapp DE, Shaw NM, Hougen HY, Agard HE, Case RM Jr, McMurry TL, Schenkman NS, Krupski TL. Effect of active versus passive void trials on time to patient discharge, urinary tract infection, and urinary retention: a randomized clinical trial. World J Urol. 2020 Sep;38(9):2247-2252. doi: 10.1007/s00345-019-03005-0. Epub 2019 Nov 15. PMID 31732771
- [Background] Wang R, Won S, Haviland MJ, Von Bargen E, Hacker MR, Li J, Lefevre R. Voiding trial outcome following pelvic floor repair without incontinence procedures. Int Urogynecol J. 2016 Aug;27(8):1215-20. doi: 10.1007/s00192-016-2975-y. Epub 2016 Feb 17. PMID 26886553
- [Background] Barr SA, Thomas A, Potter S, Melick CF, Gavard JA, McLennan MT. Incidence of successful voiding and predictors of early voiding dysfunction after retropubic sling. Int Urogynecol J. 2016 Aug;27(8):1209-14. doi: 10.1007/s00192-016-2972-1. Epub 2016 Feb 19. PMID 26894607